CLINICAL TRIAL: NCT04129411
Title: Pilot Study for the Treatment of Papillary Thyroid Carcinoma With Radiofrequency Ablation
Brief Title: Treatment of Papillary Thyroid Carcinoma With Radiofrequency Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-005486
Record Dates: First submitted 2019-10-04; First posted 2019-10-16 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2024-10

CONDITIONS: Papillary Thyroid Cancer; Papillary Thyroid Microcarcinoma
Keywords: RFA; Radiofrequency; Thyroid Cancer; Ablation techniques; Ultrasonography
MeSH Terms: conditions — Thyroid Cancer, Papillary; Papillary Thyroid Microcarcinoma; Thyroid Neoplasms

STUDY DESIGN:
Intervention Model Description: Open label single interventional series
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- RFA Group (Experimental)
  Interventions: Device: RFA

INTERVENTIONS:
Device: RFA — Radiofrequency ablation of selectively targeted thyroid nodule to treat papillary thyroid cancer.

SUMMARY:
Investigators intend to evaluate the efficiency of Radiofrequency ablation (RFA) therapy to treat papillary thyroid carcinoma.

DETAILED DESCRIPTION:
Investigators plan to identify patients with small papillary thyroid carcinoma and subject such patients to radiofrequency ablation (RFA) therapy.

Following RFA procedure patients will be monitored to study the changes in primary tumor volume, development of lymph node involvement, development of distant metastasis and changes in serum thyroid hormone levels.

Investigators will also assess the stability of these changes (need for repeat therapy) and the safety of the RFA procedure.

ELIGIBILITY:
Inclusion Criteria:

* Are adults
* Nodule with Papillary thyroid carcinoma meeting the below criteria:

  * Diagnosed by fine needle aspiration (FNA) cytology.
  * Size < 1.5 cm
  * Non-surgical therapy is considered acceptable by the treating physician
  * Radiology evaluation deems the lesion amenable to RFA therapy with minimal risk of complication

Exclusion Criteria:

* Clinical evidence for a multifocal papillary thyroid malignancy
* Clinical evidence for local or distant metastatic disease
* Pregnancy
* Vocal cord paralysis on contralateral side
* Coagulopathy or patients on anticoagulation therapy
* Patients with prior neck surgery or neck radiation
* Patients with neck anatomy that precludes easy access by RFA
* Patients with comorbidities deemed too high of a risk for general anesthesia
* Treatment with another investigational drug or intervention (within 6 weeks of planned RFA).
* Current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marius Stan, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RFA Group
Started | 5
Enrolled | 5 (Five participants were enrolled to the study.)
Completed | 5 (Five participants completed study.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Adults (18 years or older) who had Bethesda V or VI cytologic confirmation of a single-lesion small PTC (measuring less than 2 cm in largest diameter, without lymph node metastasis on neck ultrasonography) who refused standard therapy (surgical procedure or active surveillance) and underwent radiofrequency ablation. The electronic medical records of the patients were reviewed, and those without available follow-up data were excluded.
Arm/Group | RFA Group
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
Papillary Thyroid Cancer (PTC) Location [Count of Participants; unit: Participants]
  Right | 3
  Left | 2
  Isthmus | 0

OUTCOME MEASURES:

1. Primary Outcome: Changes in Thyroid Nodule Size
Description: Thyroid tumor volume shrinkage will be assessed by ultrasound and compared with pre-procedure volume (measure in mL)
Time Frame: 24 months
Population: Due to loss of follow up, some patients did not have data available at specific time interval.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | RFA Group
Number analyzed (Participants) | 5
mL
  Pre-RFA | 0.241361 (0.141814)
  3-6 months | 0.954909 (0.915872)
  7-12 months | 0.422121 (0.396916)
  13-18 months: number analyzed (Participants) | 3
  13-18 months | 0.104143 (0.076919)
  19-24 months: number analyzed (Participants) | 2
  19-24 months | 0.040035 (0.043296)

2. Secondary Outcome: Pain Related to RFA Procedure
Description: Assessed by number of participants that reported any pain related to RFA procedure
Time Frame: Up to 24 months
Population: One patient reported localized neck erythema and pain that improved within a week with over-the-counter medication.
Measure: Count of Participants; unit: Participants
Arm/Group | RFA Group
Number analyzed (Participants) | 5
Participants | 1

3. Secondary Outcome: Development of Lymph Node Involvement
Description: Assessed by the number of participants with cervical adenopathy (enlargement of lymph nodes in the neck area). Participants will be evaluated during follow-up visits.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | RFA Group
Number analyzed (Participants) | 5
Participants | 0

4. Secondary Outcome: Development of Distant Metastasis
Description: Assessed by the number of participants with distant metastasis if regional neck metastasis is detected on follow up.
Time Frame: 18 months
Population: Considering the nature of the disease, distant metastasis was not specifically evaluated if no regional neck metastasis was detected on follow up. No patients developed neck lymphadenopathy.
Measure: Count of Participants; unit: Participants
Arm/Group | RFA Group
Number analyzed (Participants) | 5
Participants | 0

5. Secondary Outcome: Safety of the RFA Procedure
Description: Assessed by the number of participants who experienced infection, hematoma, bruising, or other complications at the RFA site.
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | RFA Group
Number analyzed (Participants) | 5
Participants | 0

6. Secondary Outcome: Change in Thyroid Status
Description: Participants were tracked for thyroid status following radiofrequency ablation
Time Frame: Up to 24 months
Population: Due to loss of follow up, some patients did not have data available at specific time interval.
Measure: Count of Participants; unit: Participants
Arm/Group | RFA Group
Number analyzed (Participants) | 5
Participants
  Thyroid Status, 3-6 months: Euthyroid | 4
  Thyroid Status, 3-6 months: Hypothyroid | 0
  Thyroid Status, 3-6 months: Hyperthyroid | 1
  Thyroid Status, 3-6 months: Unknown | 0
  Thyroid Status, 7-12 months: Euthyroid | 5
  Thyroid Status, 7-12 months: Hypothyroid | 0
  Thyroid Status, 7-12 months: Hyperthyroid | 0
  Thyroid Status, 7-12 months: Unknown | 0
  Thyroid Status, 13-18 months: number analyzed (Participants) | 3
  Thyroid Status, 13-18 months: Euthyroid | 2
  Thyroid Status, 13-18 months: Hypothyroid | 0
  Thyroid Status, 13-18 months: Hyperthyroid | 0
  Thyroid Status, 13-18 months: Unknown | 1
  Thyroid Status, 19-24 months: number analyzed (Participants) | 2
  Thyroid Status, 19-24 months: Euthyroid | 2
  Thyroid Status, 19-24 months: Hypothyroid | 0
  Thyroid Status, 19-24 months: Hyperthyroid | 0
  Thyroid Status, 19-24 months: Unknown | 0

ADVERSE EVENTS:
Time Frame: 24 months
Groups:
- RFA Group: RFA: Radiofrequency ablation of selectively targeted thyroid nodule to treat papillary thyroid cancer. No adverse events were reported by participants.
Arm/Group | RFA Group
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT04129411/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT04129411/ICF_001.pdf